CLINICAL TRIAL: NCT06824688
Title: Efficacy and Safety Assessment of Single-port Versus Multi-port Robotic Surgery for Rectal Cancer: a Phase 2a Non-randomized Controlled Study Based on the IDEAL Framework
Brief Title: Single-port Versus Multi-port Robotic Surgery for Rectal Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPORTS-02
Record Dates: First submitted 2024-12-25; First posted 2025-02-13 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2024-10

CONDITIONS: Rectal Cancer Patients; Robotic Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single-port robotic total mesorectal excision (Experimental): Single-port robotic total mesorectal excision
  Interventions: Procedure: Single-port robotic total mesorectal excision
- Multi-port robotic total mesorectal excision (Active Comparator): Multi-port robotic total mesorectal excision
  Interventions: Procedure: Multi-port robotic total mesorectal excision

INTERVENTIONS:
Procedure: Single-port robotic total mesorectal excision — Single-port robotic total mesorectal excision
  Arms: Single-port robotic total mesorectal excision
Procedure: Multi-port robotic total mesorectal excision — Multi-port robotic total mesorectal excision
  Arms: Multi-port robotic total mesorectal excision

SUMMARY:
Single-port versus multi-port robotic surgery for rectal cancer

DETAILED DESCRIPTION:
This study is a phase 2a clinical trial based on the IDEAL framework, which aims to evaluate the safety and short-term clinical efficacy of single-port robotic total mesorectal excision by comparing it with multi-port robotic total mesorectal excision. The primary endpoint is short-term clinical efficacy, including intraoperative complications, blood loss, conversion rate, operation time, postoperative complications within 30 days, time to first flatus after surgery, and postoperative hospital stay. Secondary endpoints include incision length, visual analog scale (VAS) scores for postoperative pain on days 1-3, completeness of mesorectal excision grading, positive circumferential resection margin rate, positive distal resection margin rate, and the number of harvested lymph nodes.

This study was conducted in two phases:

Phase I : A single-arm study of single-port robotic radical resection for rectal cancer (n=20) Phase II : A prospective non-randomized controlled study comparing single-port (n=100) versus multi-port (n=100) robotic radical resection for rectal cancer

ELIGIBILITY:
Inclusion criteria comprised: (1) MRI-confirmed distal tumor margin <15 cm from the anal verge, (2) biopsy-proven adenocarcinoma, (3) clinical stage I-III (AJCC 8th edition) with potential downstaging post-neoadjuvant therapy, (4) intent-to-treat with sphincter preservation and primary anastomosis, (5) documented informed consent, and (6) adult patients (≥18 years).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of perioperative complications | Intraoperative and postoperative 30 days
  Perioperative complications will be described using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTACAE) v. 4.03 criteria. Complications will refer to any medical occurrence directly attributed to the surgical procedure during and within the first 30 days.
Number of participants with conversion procedures | Date of surgery (Day 1)
  The number of patients converted from robotic to open or laparoscopic surgery

SECONDARY OUTCOMES:
Pain scores | Postoperative days 1-3
  Visual Analog Scale (VAS) pain scores for patients on postoperative days 1-3
Quality of specimen | Date of surgery (Day 1)
  As proposed and published by Quirke et al（Macroscopic evaluation of rectal cancer resection specimen: clinical significance of the pathologist in quality control. J Clin Oncol. 2002 Apr 1;20(7):1729-34.）
Total length of incisions | Date of surgery (Day 1)
  Total length of all abdominal incisions (measured in millimeters).

CONTACTS AND LOCATIONS:
Overall Officials: Fan Li, Study Director — Army Medical Center (Daping Hospital), Army Medical University
Locations (1):
- Huichao Zheng, Chongqing, China